CLINICAL TRIAL: NCT00202943
Title: Comparison of Clinical Effect Between Temperature-Controlled Radio-Frequency Uvuloplasty and Laser Assisted Uvulo-Pharyngoplasty in Patients Who Snore
Brief Title: Randomized Controlled Trial of TCRFVR and LAUP in Snorers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 911007; TCVGH-917003A
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Snorer
Keywords: TCRFVR, LAUP, Snorer

INTERVENTIONS:
Procedure: TCRFVR and LAUP

SUMMARY:
We hypothesis that radiofrequency will cause less post-operative discomfort when compared with laser assited uvulopharyngoplasty. 40 patients with primary snore will be enrolled into this study. After overnight sleep test confimred that no obstructive sleep apnea existed, cases were informed consented. Then they were randomized into two groups. Post-operative pain, duration of analgesics were recorded.

DETAILED DESCRIPTION:
Although Rf group was less effective, they felt less discomfort.

ELIGIBILITY:
Inclusion Criteria:

* RDI < 5/h

Exclusion Criteria:

* Previous treated snoring, coagulation disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-03; Study Completion 2004-03

PRIMARY OUTCOMES:
LAUP is more effective in eliminating snoring

SECONDARY OUTCOMES:
However, Rf cause less post-operative discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Shih-An Liu, MD, MHA, Principal Investigator — Taichung Veterans General Hospital